CLINICAL TRIAL: NCT00556257
Title: A Pilot Randomized, Multicenter, Open-Label, Active Comparator-Controlled Trial Of A CP-690,550-Based Regimen In De Novo Kidney Allograft Recipients
Brief Title: Study Of JAK3 Inhibitor For The Prevention Of Acute Rejection In Kidney Transplant Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A3921037
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2008-05-30 (Estimated); Status verified 2008-05

CONDITIONS: Kidney Transplantation
Keywords: Immunosuppression, JAK3 inhibitor, kidney transplantation
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Arm 1 (Active Comparator): Treatment Arm 1 will also receive standard of care medications.
  Interventions: Drug: Cyclosporine
- Treatment Arm 2 (Experimental): Treatment Arm 2 will also receive select standard of care medications.
  Interventions: Drug: CP-690-,550

INTERVENTIONS:
Drug: Cyclosporine — Standard of care
  Arms: Treatment Arm 1
Drug: CP-690-,550 — CP-690550 20 mg BID in Months 1-6 then 15 mg BID in Months 7-12
  Arms: Treatment Arm 2

SUMMARY:
A new immunosuppressive drug based on the inhibition of an important enzyme in the immune system called JAK3, is being developed by Pfizer to prevent transplant rejection. In this research study, a JAK3 inhibitor or cyclosporine will be given to new kidney transplant patients for 12 months in addition to other standard transplant medications such as prednisone.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of first time kidney transplant
* Between the ages of 18 and 70 years, inclusive

Exclusion Criteria:

* Recipient of any non-kidney transplant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-08

PRIMARY OUTCOMES:
Clinical biopsy proven acute rejection rate at 6 months | 6 months

SECONDARY OUTCOMES:
Pharmacokinetics of CP-690,550 | 12 months
Lymphocyte subsets | 12 months
Posttransplant humoral alloreactivity | 12 months
Safety and tolerability of CP-690,550 | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921037&StudyName=Study%20Of%20JAK3%20Inhibitor%20For%20The%20Prevention%20Of%20Acute%20Rejection%20In%20Kidney%20Transplant%20Patients